CLINICAL TRIAL: NCT00607126
Title: Robotic Locomotor Training in Persons With Multiple Sclerosis
Brief Title: Locomotor Training in Persons With Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Barbara Giesser, Clinical Professor of Neurology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-04-064-02; RG3724-A-4 (Other: National MS Society)
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Sclerosis
Keywords: impaired ambulation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): locomotor training using body weight support on a treadmill, using robotic device to provide locomotor training. Locomotor training will be done using the Lokomat device. the patient is suspended over a treadmill while their legs are in the Lokomat, which moves the legs on the treadmill.
  Interventions: Device: Lokomat
- 2 (Active Comparator): resistive training using weights and therabands
  Interventions: Procedure: resistive training

INTERVENTIONS:
Device: Lokomat — locomotor training using body weight support on a treadmill
  Arms: 1
Procedure: resistive training — resistive training using theraband and/or weights
  Arms: 2

SUMMARY:
Locomotor training is a new exercise modality that emphasizes task specificity to promote learning and neural plasticity. It has been reported to improve walking in patients with stroke, spinal cord injury and cerebral palsy. In this study, 40 patients with impaired ambulation due to Multiple Sclerosis will be randomized to receive 36 sessions of either locomotor training or an standard resistive exercise intervention.The locomotor training will be accomplished via a robotic device, the Lokomat, which will move the patient's legs on a treadmill while they are suspended in a harness.

DETAILED DESCRIPTION:
In this study, subjects with confirmed diagnosis of Multiple Sclerosis were randomized into one of two treatment arms. Subjects in the Lokomat arm trained on the Lokomat with a supervising physical therapist for 20-30 minutes/session 3 times/week. The Lokomat is a robotic exoskeleton which enables the subject to step on a moving treadmill. Subjects were suspended in a harness while in the Lokomat with full to partial body weight support as needed. After the training in the Lokomat, they practiced overground walking for 10 minutes.

The other treatment arm had subjects engage in resistance training with weights and resistance elastic bands matched to the Lokomat group for intensity, duration and frequency. they did not practice overground walking.

Primary outcome measure was speed to accomplish 25' timed walk.

ELIGIBILITY:
Inclusion Criteria:

* Persons with Secondary progressive or Primary Progressive Multiple Sclerosis who are ambulatory with difficulty and /or assistive device

Exclusion Criteria:

* Ataxia
* Unable to ambulate
* Within 3 months of exacerbation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara S Giesser, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giesser B, Beres-Jones J, Budovitch A, Herlihy E, Harkema S. Locomotor training using body weight support on a treadmill improves mobility in persons with multiple sclerosis: a pilot study. Mult Scler. 2007 Mar;13(2):224-31. doi: 10.1177/1352458506070663. PMID 17450642
- [Background] Giesser B, Herlihy E, Plummer D'Amato P et al. Randomized controlled trial of robotic locomotor training in persons with MS. Multiple Sclerosis Journal 17S481 ( 2011)
- [Result] Giesser B, Herlihy, E, PlummerD'Amato P, et al. Locomotor training may improve cognitive performance in persons with MS. Neurology 72 ( Suppl.3) A 405 (2009)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective subjects were recruited from the MS clinic population of the UCLA Dep't/ of Neurology and from the general MS population in Los Angeles between 2007-2009. Recruitment flyers were approved by the UCLA Institutional Review board.
Pre-assignment Details: 38 subjects were consented and randomized; two subjects volitionally dropped out before participating in the study; this accounts for the discrepancy..
Groups:
- Lokomat Training Using Body Weight Support on a Treadmill: Locomotor training using body weight support on a treadmill, using robotic device to provide locomotor training. Locomotor training will be done using the Lokomat device. The Lokomat device is a robotic exoskeleton which fits over the patient's legs while they are suspended in a harness over a standard treadmill. the patient is suspended over a treadmill while their legs are in the Lokomat, which moves the legs on the treadmill. Patient had to be ambulatory with or without an assistive device. The amount of body weight support is gradually increased or decreased as needed.Partients were also given feedback by the physical therapist while they were walking on the treadmill. Patients trained for 30-40 minutes per session, for 3X/week. The average speed of training was 2.4km.hr. After lokomat training, the patients practiced over ground walking with the therapist for 15 minutes after each session.
- Resistive Training: resistive training using weights and therabands
  This group trained for the same amount of time as the Lokomat group, i.e.3X/week for 30-40 minutes per session. they used resistive weights and /or theraband resistive bands to accomplish training. Exercises were done in supine, lying sitting and standing positions. Large muscle groups in both upper and lower extremities were trained. Patients completed 3 sets of 8-12 reps of each exercise, and performed 8-10 different exercises in each session.
Period: Overall Study
Arm/Group | Lokomat Training Using Body Weight Support on a Treadmill | Resistive Training
Started | 17 | 19
Completed | 17 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lokomat Training Using Body Weight Support on a Treadmill | Resistive Training | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36
EDSS [Mean (Full Range); unit: units on a scale] — this is a scale which measures disability. each participant will have their own individual EDSS. The EDSS is the abbreviation for the Expanded Disability Status Scale. It is scored from information obtained the neurologic exam and goes from 0-10. O is "normal "and 10 is "dead". A higher number therefore connotes worse physical disability.
  units on a scale | 6.5 [5.5 to 6.5] | 6.0 [5 to 6.5] | 6.3 [5 to 6.5]

OUTCOME MEASURES:

1. Primary Outcome: Walking Speed as Assessed by 25' Timed Walk
Description: This is the time needed for participant to walk 25 feet. Participant walks on a level surface. the walk from start to finish is timed with a stop watch three measures are done and the average value is entered.
Time Frame: at beginning,mid point, end and 12 weeks after intervention
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Lokomat Training Using Body Weight Support on a Treadmill | Resistive Training
Number analyzed (Participants) | 17 | 19
seconds
  25"TW baseline | 22.7 (17.6) | 10.6 (4.9)
  25'TW midpoint | 23.9 (20.9) | 9.8 (4.3)
  25'TW end point | 19.4 (15.2) | 9.6 (3.7)
  25'TW post | 21.7 (16.7) | 10.5 (4.3)

2. Secondary Outcome: Distance
Description: distance assessed by 6 minute walk test
Time Frame: baseline, mid point, end and 12 weeks after training
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Lokomat Training Using Body Weight Support on a Treadmill | Resistive Training
Number analyzed (Participants) | 17 | 19
feet
  6 min walk baseline | 367 (241) | 753 (232.3)
  6 min walk midpoint | 474 (354) | 813 (253.8)
  6 minute walk end point | 436 (288) | 769 (261.9)
  6 minute walk post | 457 (300.5) | 742 (248.2)

3. Secondary Outcome: Fatigue
Description: fatigue assessed by modified fatigue impact scale. This is a 21 item questionnaire which has a range from 0-84. Higher scores indicate more impact of fatigue on physical and cognitive functioning.
Time Frame: baseline, mid, completetion, 3 months post
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lokomat Training Using Body Weight Support on a Treadmill | Resistive Training
Number analyzed (Participants) | 17 | 19
units on a scale
  MFIS baseline | 34.1 (14.1) | 37.7 (15.6)
  MFIS mid point | 26.7 (13.7) | 29.4 (15.0)
  MFIS end point | 26.8 (16.6) | 29.9 (17.7)
  MFIS post | 27.4 (19.8) | 35.3 (15.9)

4. Secondary Outcome: PASAT
Description: Cognitive measure of attention and information processing speed. Score goes from 0-60 with higher number indicating better performance. Scores are expressed as mean chamge rfom baseline; negative numbers indicate worse performance
Time Frame: baseline, mid, completion, 3 months post training
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lokomat Training Using Body Weight Support on a Treadmill | Resistive Training
Number analyzed (Participants) | 17 | 19
units on a scale
  PASAT baseline | 48.2 (5.1) | 46.8 (3.8)
  PASAT Mid point | 0.06 (1.17) | 0.42 (1.03)
  PASAT end point | 1.3 (1.13) | 0.58 (1.03)
  PASAT post | 1.90 (1.13) | -0.91 (1.13)

ADVERSE EVENTS:
Arm/Group | Lokomat Training Using Body Weight Support on a Treadmill | Resistive Training
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 0/19

LIMITATIONS AND CAVEATS:
This was a small study and the number of subjects enrolled may not have been sufficient to show an effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No